CLINICAL TRIAL: NCT01255774
Title: Serial Retinal Thickness Changes And Scotoma Size Measured With Lucentis Therapy Measured Using The Optical Coherence Tomography (OCT) Scanning Laser Ophthalmoscope (SLO) And The Foresee Preferential Hyperacuity Perimeter
Brief Title: Serial Retinal Thickness Changes And Scotoma Size Measured With Lucentis Therapy
Acronym: FVF4193s
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Richard Rosen, MD, Vice Chairman of Dept of Ophthalmology and Director of Research, New York Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYEE-07.14
Record Dates: First submitted 2010-12-04; First posted 2010-12-07 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Age Related Macular Degeneration
Keywords: subfoveal CNV; Wet (Exudative) AMD; macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental): Open Label use of Ranibizumab for wet age related macular degeneration
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — An open-label, study of intravitreally administered ranibizumab
  Other Names: Lucentis

SUMMARY:
The rationale for evaluating LucentisTM (a recombinant humanized anti-human Vascular Endothelial Growth Factor (VEGF) monoclonal antibody (Fab) in patients with neovascular (wet) Age related Macular Degeneration (AMD) is based on the strong correlation between VEGF levels in aqueous and vitreous humor and active blood vessel formation. LucentisTM has been shown to maintain or improve vision in wet AMD. Since the treatments do not halt the loss of visual acuity in wet AMD, it is important to accurately measure anatomic response to treatments thereby enhancing the ability to understand patterns of response and predict the necessity for continued therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Subjects of either gender, Age > 50 years
* Best corrected visual acuity in the study eye between 20/40 and 20/320.
* Subfoveal choroidal neovascularization, secondary to age related macular degeneration.
* Any subretinal hemorrhage must comprise no more than 50% of total lesion size.
* Clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography
* Men must use barrier contraception or abstinence throughout the study.
* Ability to return for all study visits

Exclusion Criteria:

* Had ocular surgery within the past 60 days in the study eye.
* Had previous refractive eye surgery (RK, PRK, LASIK, ALK, etc.) within the past 3 months for the study eye.
* Has intraocular pressure ≥ 25 mmHg in the study eye.
* Has posterior uveitis in the study eye.
* Has ongoing infection in the study eye.
* Has retinal or optic nerve disease that could independently affect visual acuity including high axial myopia (>-8.00 D) and diabetic retinopathy in the study eye.
* Has anterior segment and vitreous abnormalities that would preclude adequate observation of the fundus for photographs and fluorescein angiography in the study eye.
* Has received investigational therapy within 60 days prior to study entry.
* Has been previously enrolled in or previous treatment with MSI-1256F for injection.
* Has received prior approved treatment for subfoveal CNV within 60 days to study entry.
* Has clinically uncontrolled diabetes mellitus.
* Has other condition the investigator considers to be sound reasons for exclusion (e.g., lack of motivation, history of poor compliance, concomitant illnesses, personality disorder, mental condition, drug abuse, use of neuroleptics, physical or social condition predicting difficulty in long-term follow-up).
* Has an allergy to sodium fluorescein dye.
* Currently uses systemic or topical medications known to be toxic to the retina, lens, or optic nerve, such as deferoxamine, chloroquine/hydrochloroquine, tamoxifen, chlorpromazine, phenothiazines, steroids and ethambutol.
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.

Ages: 51 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Central retinal thickness | 12 months
  To measure the mean change in central retinal thickness as measured by OCT/ SLO and Stratus OCT from Baseline to Month 12.

SECONDARY OUTCOMES:
change in central scotoma lesion size, density and distortion due to neovascularization | 12 months
  To measure the mean change in central scotoma lesion size and density as measured on OCT/ SLO microperimeter from Baseline to Month 12.
  To measure the mean change in the scotoma size and distortion due to neovascularization as measured on the PHP from Baseline to Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Rosen, MD, Principal Investigator — New York Eye and Ear Infirmary
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States